CLINICAL TRIAL: NCT05106972
Title: A Single Center, Prospective Study of Umbilical Cord Mesenchymal Stem Cell Transplantation for Decompensated Hepatitis B Cirrhosis
Brief Title: Umbilical Cord Mesenchymal Stem Cell Transplantation for Decompensated Hepatitis B Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asia Stem Cell Regenerative Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT20181032
Record Dates: First submitted 2021-09-19; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UC-MSC infusion (Experimental): UC-MSC infusion by intravenus, 1*10^8 cells/dose, 2 doses (apart from 24weeks)
  Interventions: Drug: UC-MSC infusion

INTERVENTIONS:
Drug: UC-MSC infusion — UC-MSC infusion by introvenus

SUMMARY:
This study aims to evaluate the safety and clinical efficacy of umbilical cord mesenchymal stem cell transplantation for decompensated hepatitis B cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 60 (male or female)
* Diagnosed chronic decompensated hepatitis B cirrhosis with a course of more than 5 years
* Not suitable for liver transplantation or there is no donor liver source
* No serious bleeding tendency or active bleeding
* No hepatic encephalopathy
* After strict medical conservative treatment for more than 6 months, there was no relief of symptoms or significant improvement of quality of life score
* Subjects voluntarily participate in this study and sign informed consent

Exclusion Criteria:

* Be less than 20 years old or more than 60 years old
* Cirrhosis caused by other causes such as alcoholic hepatitis, hepatitis C virus and autoimmune hepatitis
* Found liver malignant tumor or the family history of liver malignant tumor in the third generation of their direct relatives
* Patients with hypersplenism who need splenectomy
* History of tumors in other organs
* PT prolongation is greater than 3 seconds
* Use of human serum albumin within 3 weeks prior to clinical registration
* Clinically significant upper gastrointestinal bleeding events occurred within 4 weeks before clinical registration
* Spontaneous peritonitis
* Active infection (viral or bacterial)
* Pregnant or lactating women
* The researcher considers it inappropriate to participate in this study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with abnormal Total bilirubin | Changes from baseline to 72 weeks
Number of Participants with abnormal albumin | Changes from baseline to 72 weeks
Ishak Inflammation Rating System | Changes from baseline to 72 weeks
Ishak Fibrosis Score | Changes from baseline to 72 weeks

SECONDARY OUTCOMES:
Overall survival (OS) | Changes from baseline to 72 weeks
HBV-DNA | Changes from baseline to 72 weeks
incidence of liver cancer | Changes from baseline to 72 weeks
Number of Participants with abnormal immunoglobulin | Changes from baseline to 72 weeks
portal vein flow rate | Changes from baseline to 72 weeks
portal vein width | Changes from baseline to 72 weeks
abdominal volume | Changes from baseline to 72 weeks
Number of Participants with abnormal coagulation function | Changes from baseline to 72 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Haikou People's Hospital, Haikou, China

IPD SHARING:
Plan to Share IPD: Undecided